CLINICAL TRIAL: NCT04720417
Title: A Phase II Trial of Defactinib (VS-6063) Combined With VS-6766 (CH5126766) in Patients With Metastatic Uveal Melanoma
Brief Title: Defactinib and VS-6766 for the Treatment of Patients With Metastatic Uveal Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial enrollment was stopped early by study sponsors (before the anticipated accrual of 18 patients) due to no patients having significant reduction in disease.
Sponsor: Thomas Jefferson University (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20P.1113; JT 16166 (Other: JeffTrial Number)
Record Dates: First submitted 2020-12-07; First posted 2021-01-22 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — benzamide; defactinib; RO5126766; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (defactinib, VS-6766) (Experimental): Patients receive defactinib PO BID and VS-6766 PO BIW (Monday and Thursday or Tuesday and Friday) for 3 weeks in every cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Defactinib Hydrochloride; Drug: Raf/MEK Inhibitor VS-6766; Procedure: Biopsy

INTERVENTIONS:
Drug: Defactinib Hydrochloride — Given PO
  Other Names: 1073160-26-5; Benzamide; N-methyl-4-((4-(((3-(methyl(methylsulfonyl)amino)-2-pyrazinyl)methyl)amino)-5-(trifluoromethyl)-2-pyrimidinyl)amino)-Hydrochloride (1:1); PF-04554878; VS-6063
Drug: Raf/MEK Inhibitor VS-6766 — Given PO
  Other Names: CH5126766; 946128-88-7; CH-5126766; CKI-27; R-7304; RG 7304; RG-7304; RO-5126766 FREE BASE; RO5126766; VS 6766; VS-6766; AVUTOMETINIB
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase II trial studies the effect of combining defactinib and VS-6766 in treating patients with uveal melanoma that has spread to other places in the body (metastatic). The way cells communicate with one another (different cell signaling pathways) are overactive in uveal melanoma tumor cells. Giving defactinib together with VS-6766 may block pathways that are important for the growth of uveal melanoma cells, and may result in shrinkage or stabilization of the cancer and prolonged time to disease progression and survival.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To investigate the potential efficacy of the combination of defactinib hydrochloride (defactinib [VS-6063]) and Raf/MEK serine/threonine kinase inhibitor RO5126766 (VS-6766) in patients with metastatic uveal melanoma.

SECONDARY OBJECTIVES:

I. To assess the effectiveness of defactinib in combination with VS-6766 in patients with metastatic uveal melanoma (MUM).

II. To assess the safety and toxicity profile of the combination of defactinib and VS6766.

EXPLORATORY OBJECTIVES:

I. To study the pharmacodynamic profile of defactinib in combination with VS-6766 in pre-treatment, on-treatment, and post-treatment tumor biopsies.

II. To investigate mechanisms of resistance to the combination of defactinib and VS-6766.

III. To investigate the potential efficacy of circulating cell free deoxyribonucleic acid (DNA) for prediction/monitoring.

OUTLINE:

Patients receive defactinib orally (PO) twice daily (BID) and VS-6766 PO twice a week (BIW) (Monday and Thursday or Tuesday and Friday) for 3 weeks in every cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy at baseline, after cycle 1 or 2, and post-treatment.

After completion of study treatment, patients are followed every 3 months until death or up to 2 years after the last patient is enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic uveal melanoma
* Predicted life expectancy of at least 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 based on spiral computed tomography (CT) or magnetic resonance imaging (MRI) scan, all radiology studies must be performed within 28 days prior to registration. Corrected QT interval (QTc) < 470 ms (as calculated by the Fridericia correction formula, averaged over 3 electrocardiograms [ECGs])
* Hemoglobin (Hb) >= 9.0 g/dL (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Platelet count >= 100 x 10^9/L (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Serum bilirubin =< 1.5 x upper limit of normal (ULN) (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Albumin >= 3.0 mg/dL (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Creatine phosphokinase (CPK) =< 2.5 x ULN (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 2.5 x ULN unless raised due to tumor in which case up to 5 x ULN is permissible (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Calculated creatinine clearance >= 45 mL/min by the Cockcroft-Gault formula (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* International normalized ratio (INR) =< 1.5 in absence of anticoagulation or therapeutic levels in presence of anticoagulation (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Partial thromboplastin time (PTT) =< 1.5 x ULN in absence of anticoagulation or therapeutic levels in presence of anticoagulation (performed within two weeks [day -14 to day 1] before the patient goes on the trial)
* Patients with adequate cardiac function (left ventricular ejection fraction >= 50%) by echocardiography or multigated acquisition scan (MUGA) scan
* No active retinopathy or retinal vein occlusion confirmed by full ophthalmological exam in the eye unaffected by uveal melanoma
* Adequate recovery from toxicities related to prior treatments to at least grade 1 by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Exceptions include alopecia and peripheral neuropathy grade =< 2. Subjects with other toxicities that are stable on supportive therapy may be allowed to participate with prior approval by the sponsor
* Men and women aged 18 years or over
* Females with reproductive potential and their male partners agree to use highly effective method of contraceptive (per Clinical Trial Facilitation Group [CFTG] recommendations during the trial and for 3 months following the last dose of study drug)
* Written (signed and dated) informed consent and be capable of cooperating with treatment and follow-up
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Exclusion Criteria:

1. Radiotherapy (except for palliative reasons), endocrine therapy, biological therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) before treatment.
2. Ongoing toxic manifestations of previous treatments. Exceptions to this are alopecia or certain Grade 1 toxicities, which in the opinion of the Investigator and the DDU should not exclude the patient.
3. Known untreated or active central nervous system (CNS) metastases (progressing or requiring corticosteroids for symptomatic control). Patients with a history of treated CNS metastases are eligible, provided they meet all of the following criteria:

   * Evaluable or measurable disease outside the CNS is present.
   * Radiographic demonstration of improvement upon the completion of CNS- directed therapy and no evidence of interim progression between the completion of CNS- directed therapy and the baseline disease assessment for at least 28 days.
4. Gilbert syndrome diagnosed with elevated indirect (unconjugated) bilirubin ( >1.2 mg/dl) at least two occasions with normal direct bilirubin in the absence of hemolysis or structural liver damage.
5. Ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum or urine pregnancy test before enrollment and agree to use two medically approved forms of contraception (oral, injected or implanted hormonal contraception and condom, have an intra-uterine device and condom, diaphragm with spermicidal gel and condom) from time of consent, during the trial and for six months afterwards are considered eligible.
6. Male patients with partners of child-bearing potential (unless they agree to take measures not to father children by using one form of medically approved contraception [condom plus spermicide] during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (for example, condom plus spermicidal gel) to prevent exposure to the fetus or neonate.
7. Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study and from which the patient has not yet recovered.
8. Treatment with warfarin. Patients on warfarin for DVT/PE can be converted to low-molecular-weight heparin (LMWH).
9. Acute or chronic pancreatitis.
10. At high medical risk because of non-malignant systemic disease including active uncontrolled infection.
11. Known to be serologically positive for hepatitis B, hepatitis C or human immunodeficiency virus (HIV).
12. Patients with the inability to swallow oral medications or impaired gastrointestinal absorption due to gastrectomy or active inflammatory bowel disease.
13. History of abdominal fistula, gastro-intestinal perforation, or diverticulitis.
14. Patients with history of symptomatic cholelithiasis or cholecystitis within six months before enrollment.
15. Concurrent ocular disorders in the eye unaffected by uveal melanoma:

    1. Patients with history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes
    2. Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    3. Patients with a history of corneal erosion (instability of corneal epithelium), corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions.
16. Concurrent congestive heart failure, prior history of class III/ IV cardiac disease (New York Heart Association [NYHA]), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
17. Patients exposed to strong CYP3A4 and strong CYP2C9 inhibitors within 7 days prior to the first dose. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information.
18. Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this Phase II study of VS-6766 in combination with VS-

6063. Participation in an observational trial would be acceptable. 19. Patients with a history of hypersensitivity to any of the inactive ingredients (hydroxypropylmethylcellulose, mannitol, magnesium stearate) of the investigational product. 20. Prior corticosteroids as anti-cancer therapy within a minimum of 14 days of first receipt of study drugs. 21. Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rino Seedor, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramms DJ, Raimondi F, Arang N, Herberg FW, Taylor SS, Gutkind JS. Galphas-Protein Kinase A (PKA) Pathway Signalopathies: The Emerging Genetic Landscape and Therapeutic Potential of Human Diseases Driven by Aberrant Galphas-PKA Signaling. Pharmacol Rev. 2021 Oct;73(4):155-197. doi: 10.1124/pharmrev.120.000269. PMID 34663687

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject did not initiate treatment due to rapid disease progression.
Period: Overall Study
Arm/Group | Treatment (Defactinib, VS-6766)
Started | 13
Completed | 12
Not Completed | 1
Not completed — one subject did not initiate treatment due to rapid disease progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Defined as complete response (CR) + partial response (PR) + stable disease (SD) and determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Time Frame: From baseline through last follow-up visit (up to 24 months per participant)
Population: No subjects met this criteria. The trial was closed before the anticipated accrual of 18 patients, but of the 12 patients that were treated the best overall response rate was 0% as no patient achieved CR or PR. All subjects died or relapsed disease/progression and did not complete.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 12
Participants | 0

2. Primary Outcome: Disease Control Rate
Description: Defined as CR+PR+SD and determined by RECIST criteria version 1.1. All estimates of rates will be presented with corresponding 95% exact confidence intervals. For disease control rates, the method of Atkinson and Brown will be used to allow for the two-stage design.
Time Frame: From baseline through last follow-up visit (up to 24 months per participant)
Population: The trial was closed before the anticipated accrual of 18 patients, but of the 12 patients that were treated the disease control rate was 50% (6 patients with SD).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 12
Participants | 6

3. Secondary Outcome: Progression-free Survival (PFS)
Description: A Kaplan Meier graph and median PFS will be presented overall and by cohort.
Time Frame: From first dose of study drug until disease progression or death (whichever occurs first). Up to 24 months per participant.
Population: 12 patients received at least one dose of study drug and were included in progression-free survival (PFS) and follow-up analysis population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 12
Months
  Progression-Free Survival | 3.04 [1.91 to 6.15]
  Follow up period | 20 [6.77 to 26.8]

4. Secondary Outcome: Overall Survival (OS)
Description: A Kaplan Meier graph will be presented overall and by cohort.
Time Frame: From first dose of study drug until disease progression or death (whichever occurs first). Up to 14 months.
Population: Trial closed prematurely based on limited clinical activity as reflected by the low rate of short-lasting disease control without any partial responses, slow enrollment, and the heavily pretreated study population reflecting the changing treatment landscape.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 12
Participants | 2

5. Secondary Outcome: Incidence of Adverse Events
Description: Will determine causality of each adverse event to defactinib and VS-6766 and grading severity according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Estimates of toxicity rates will be presented with corresponding 95% exact confidence intervals. Safety variables will be summarized by descriptive statistics. Laboratory variables will be described using the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Adverse events (AEs) will be reported for each dose level and presented as tables of frequency of AEs by body system and by worse severity grade observed.
Time Frame: From baseline through last follow-up visit (up to 14 months)
Measure: Number; unit: Number of AEs
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 12
Number of AEs | 43

6. Other Pre Specified Outcome: Changes in Tumor Metabolic Activity
Description: Tumor samples will be analyzed for changes in tumor metabolic activity.
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: Analysis not performed. Trial closed prematurely based on limited clinical activity as reflected by the low rate of short-lasting disease control without any partial responses, slow enrollment, and the heavily pretreated study population reflecting the changing treatment landscape.
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

7. Other Pre Specified Outcome: Changes in Signaling to the ERK Pathways
Description: Tumor samples will be analyzed for changes in signaling to the ERK pathways. Subjects grouped (Progressive Disease v Stable Disease) for sake of results reporting.
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: 4 total patients with pre- and post- biopsy samples were available. Pre- vs post- biopsy samples was assessed for changes in active ERK (pERK)
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Defactinib, VS-6766) - Subjects With Progressive Disease; Treatment (Defactinib, VS-6766) - Subjects With Stable Disease: Patients receive defactinib PO BID and VS-6766 PO BIW (Monday and Thursday or Tuesday and Friday) for 3 weeks in every cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Defactinib Hydrochloride: Given PO
  Raf/MEK Inhibitor VS-6766: Given PO
  Biopsy: Undergo tumor biopsy
Arm/Group | Treatment (Defactinib, VS-6766) - Subjects With Progressive Disease | Treatment (Defactinib, VS-6766) - Subjects With Stable Disease
Number analyzed (Participants) | 2 | 2
Participants
  Reduction in active ERK (pERK) | 0 | 2
  No change in active ERK (pERK) | 2 | 0

8. Other Pre Specified Outcome: Changes in Cell Proliferation (Ki67)
Description: Tumor samples will be analyzed for changes in cell proliferation
Time Frame: Baseline up to 2 years after the last patient is enrolled
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Changes in Apoptosis Induction (Caspase Activation)
Description: Tumor samples will be analyzed for changes in apoptosis induction
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Changes in Tumor Microenvironment
Description: Tumor samples will be analyzed for changes in tumor microenvironment
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Detection of Biomarkers of Resistance
Description: Tumor samples will be analyzed. The specific type and number of biomarkers from the tumor samples will be decided during the course of the study and documented in the study records.
Time Frame: Up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Circulating Free Deoxyribonucleic Acid (DNA)
Description: Will correlate circulating free DNA with cancer remission and predicting cancer relapse.
Time Frame: Up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Changes in Signaling to the YAP Pathways
Description: Tumor samples will be analyzed for changes in signaling to the YAP pathways
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Changes in Signaling to the FAK Pathways
Description: Tumor samples will be analyzed for changes in signaling to the FAK pathways
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Changes in Signaling to the PI3K TOR Pathways
Description: Tumor samples will be analyzed for changes in signaling to the PI3K TOR pathways
Time Frame: Baseline up to 28 days after the last dose of treatment
Population: as for outcome 6
Arm/Group | Treatment (Defactinib, VS-6766)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From first dose to 28 days after last dose of study drug (approximately 3-14 months)
Description: Adverse events (serious and non-serious) were collected from time of informed consent to 28 days after last dose of study drug.
Arm/Group | Treatment (Defactinib, VS-6766)
All-Cause Mortality (participants affected / at risk) | 11/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Defactinib, VS-6766) (N=12)
Skin Infection - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1) — Not related to study drug. Resulted from trauma to the area after MVA (motor vehicle accident)
Hip dislocation - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated [The adverse event (toxicity) is not related to the investigational agent(s).]
CPK Increased - Grade 3 (Investigations) | 1 (1)
GGT increased - Grade 3 (Hepatobiliary disorders) | 1 (1)
Hypokalemia - Grade 3 (Metabolism and nutrition disorders) | 1 (1)
Syncope - Grade 3 (Nervous system disorders) | 1 (1)
Urticaria - Grade 3 (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Defactinib, VS-6766) (N=12)
Abdominal bloating - Grade 1 (Gastrointestinal disorders) | 1 (1)
Acneiform rash - Grade 1 (Skin and subcutaneous tissue disorders) | 12 (18)
Acneiform rash - Grade 2 (Skin and subcutaneous tissue disorders) | 4 (4)
Alopecia - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (2)
Alopecia - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Blurred Vision - Grade 1 (Eye disorders) | 6 (9)
Concentration impairment - Grade 1 (Nervous system disorders) | 1 (1)
Constipation - Grade 1 (Gastrointestinal disorders) | 2 (2)
CPK increased - Grade 1 (Investigations) | 1 (1)
CPK increased - Grade 2 (Investigations) | 1 (1)
Diarrhea - Grade 1 (Gastrointestinal disorders) | 8 (11)
Diarrhea - Grade 2 (Gastrointestinal disorders) | 1 (1)
Dizziness - Grade 1 (Nervous system disorders) | 5 (5)
Dry Mouth - Grade 1 (Gastrointestinal disorders) | 3 (4)
Dry Skin - Grade 1 (Skin and subcutaneous tissue disorders) | 5 (7)
Dysgeusia - Grade 1 (Nervous system disorders) | 3 (3)
Edema - Limbs - Grade 1 (General disorders) | 5 (8)
Edema - Limbs - Grade 2 (General disorders) | 1 (1)
Fatigue - Grade 1 (General disorders) | 8 (8)
Fatigue - Grade 2 (General disorders) | 1 (1)
Fever - Grade 1 (General disorders) | 3 (3)
Fever - Grade 2 (General disorders) | 1 (1)
GERD - Grade 1 (Gastrointestinal disorders) | 4 (4)
GGT increased - Grade 1 (Hepatobiliary disorders) | 1 (1)
Hoarseness - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Maculopapular rash - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Mucositis oral/stomatitis - Grade 1 (Gastrointestinal disorders) | 4 (4)
Nausea - Grade 1 (Gastrointestinal disorders) | 8 (8)
Night Sweats - Grade 1 (Skin and subcutaneous tissue disorders) | 2 (2)
PICA - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Platelet count decreased - Grade 1 (Blood and lymphatic system disorders) | 1 (1)
Pocket of subfoveal fluid right eye - Grade 1 (Eye disorders) | 1 (1)
Maculopapular Rash - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
Thrush - Grade 1 (Gastrointestinal disorders) | 1 (1)
Thrush - Grade 2 (Gastrointestinal disorders) | 1 (1)
Vomiting - Grade 1 (Gastrointestinal disorders) | 3 (3)
Abdominal pain - Grade 1 (Gastrointestinal disorders) | 5 (6)
Adrenal insufficiency - Grade 1 (Endocrine disorders) | 1 (1)
Alanine aminotransferase increased - Grade 1 (Hepatobiliary disorders) | 1 (1)
Allergic Rhinitis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anorexia - Grade 1 (Metabolism and nutrition disorders) | 2 (3)
Anxiety - Grade 1 (Psychiatric disorders) | 5 (5)
Anxiety - Grade 2 (Psychiatric disorders) | 2 (2)
Arthralgia - Grade 1 (Musculoskeletal and connective tissue disorders) | 5 (6)
Arthralgia - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Ascites - Grade 1 (Gastrointestinal disorders) | 1 (1)
Ascites - Grade 2 (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased - Grade 1 (Hepatobiliary disorders) | 1 (1)
Back Pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (3)
Back Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Bilateral Myopia - Grade 1 (Eye disorders) | 1 (1)
Bone Spur - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Pain - Grade 2 (Reproductive system and breast disorders) | 1 (1)
Broken nail - left thumb - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising - Grade 1 (Injury, poisoning and procedural complications) | 1 (2)
Burning sensation - Back - Grade 1 (Nervous system disorders) | 1 (1)
Cataract - Grade 1 (Eye disorders) | 2 (2)
Chills - Grade 1 (General disorders) | 2 (2)
Cholesterol high - Grade 1 (Investigations) | 2 (2)
Cholesterol high - Grade 2 (Investigations) | 1 (1)
Cognitive Disturbance - Grade 1 (Nervous system disorders) | 2 (2)
Cough - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cystoid Macular Edema - Grade 2 (Eye disorders) | 1 (1)
Depression - Grade 1 (Psychiatric disorders) | 3 (3)
Dry Eye - Grade 1 (Eye disorders) | 1 (1)
Duodenal Ulcer - Grade 1 (Gastrointestinal disorders) | 1 (1)
Ear Pain - Grade 1 (Ear and labyrinth disorders) | 1 (1)
Edema - Trunk - Grade 1 (General disorders) | 1 (1)
Fall - Grade 1 (Injury, poisoning and procedural complications) | 2 (2)
Fall - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Fracture - Grade 2 (Injury, poisoning and procedural complications) | 1 (1)
Gait Disturbance - Grade 1 (General disorders) | 1 (2)
Gait Disturbance - Grade 2 (General disorders) | 1 (2)
Gastritis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Gastroparesis - Grade 1 (Gastrointestinal disorders) | 1 (1)
Genital edema - Grade 1 (Reproductive system and breast disorders) | 1 (1)
Glaucoma - Grade 1 (Eye disorders) | 1 (1)
Headache - Grade 1 (Nervous system disorders) | 4 (5)
Headache - Grade 2 (Nervous system disorders) | 1 (1)
Heart Murmur - Grade 1 (Cardiac disorders) | 2 (2)
Hematoma - Grade 1 (Vascular disorders) | 1 (1)
Herpes simplex reactivation - Grade 1 (Infections and infestations) | 1 (1)
Hip Dislocation - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (2)
Hypertension - Grade 1 (Vascular disorders) | 2 (2)
Hypokalemia - Grade 1 (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia - Grade 2 (Metabolism and nutrition disorders) | 1 (1)
Hypotension - Grade 1 (Vascular disorders) | 1 (1)
Hypothyroidism - Grade 1 (Endocrine disorders) | 4 (4)
Hypothyroidism - Grade 2 (Endocrine disorders) | 1 (1)
Injection site reaction - Grade 1 (Injury, poisoning and procedural complications) | 1 (1)
Insomnia - Grade 1 (Psychiatric disorders) | 4 (4)
Hereditary Hemochromatosis (Congenital, familial and genetic disorders) | 1 (1)
Joint Pain - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Left shoulder nodule - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Localized edema - Grade 1 (General disorders) | 1 (2)
mitral regurgitation - Grade 2 (Cardiac disorders) | 1 (1)
Mouth Sores - intermittent - Grade 1 (Gastrointestinal disorders) | 1 (1)
Muscle Cramp - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Nail Infection - Grade 1 (Infections and infestations) | 1 (1)
Nail Loss - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal congestion - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Neck pain - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Nocturia - Grade 1 (Renal and urinary disorders) | 3 (3)
Pain - Hip - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Hip - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (2)
Pain - Muscle Soreness - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - Shoulder - Grade 1 (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain - Shoulder - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Paronychia - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral sensory neuropathy - Grade 1 (Nervous system disorders) | 1 (1)
Postnasal drip - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritus - Grade 1 (Skin and subcutaneous tissue disorders) | 4 (4)
Pulmonary nodules - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal perforation - Grade 1 (Gastrointestinal disorders) | 2 (2)
Scalp Pain - Grade 1 (Skin and subcutaneous tissue disorders) | 3 (3)
Scalp Pain - Grade 2 (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus bradycardia - Grade 1 (Cardiac disorders) | 2 (2)
Sinusitis - Grade 2 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin abrasion - hand - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin discoloration - eye lid - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection - Grade 2 (Infections and infestations) | 1 (1)
Skin lacerations - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Sleep Apnea - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1)
sore bump on left shoulder - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Spinal Fracture - Grade 2 (Musculoskeletal and connective tissue disorders) | 1 (1)
Stomach Pain - Grade 1 (Gastrointestinal disorders) | 1 (1)
Strain (foot) - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1)
Stye - Grade 1 (Eye disorders) | 1 (1)
subcutaneous tumor removal - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)
Tremor - Grade 2 (Nervous system disorders) | 1 (1)
Tumor Pain - Grade 1 (General disorders) | 1 (1)
Upper respiratory infection - Grade 2 (Infections and infestations) | 1 (1)
Ureteral Polyps - Grade 1 (Renal and urinary disorders) | 1 (1)
Urinary tract infection - Grade 2 (Infections and infestations) | 2 (2)
Urticaria - Grade 1 (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/17/NCT04720417/Prot_SAP_000.pdf